CLINICAL TRIAL: NCT06996184
Title: A Phase 1, Randomized, Open-label Study to Characterize the Effect of Food on the Oral Bioavailability of a Prolonged-release Formulation of Vamifeport in Healthy Adult Subjects
Brief Title: Effect of Food on the Oral Bioavailability of a Prolonged-release Formulation of Vamifeport in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CSL624_1006
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1: Vamifeport Fasted then Fed (Experimental): In sequence 1, eligible participants assigned to sequence 1 will receive a single vamifeport dose on an empty stomach on Day 1 (fasted condition), undergo a washout period, and then receive a single vamifeport dose after a standardized high-fat meal (fed condition) on Day 6.
  Interventions: Drug: Vamifeport (PR formulation)
- Sequence 2: Vamifeport Fed then Fasted (Experimental): In sequence 2, eligible participants assigned to sequence 2 will receive a single vamifeport dose after a standardized high-fat meal on Day 1 (fed condition), undergo a washout period, and then receive a single vamifeport dose on an empty stomach (fasted condition) on Day 6.
  Interventions: Drug: Vamifeport (PR formulation)

INTERVENTIONS:
Drug: Vamifeport (PR formulation) — Vamifeport will be administered orally
  Other Names: CSL624

SUMMARY:
This is a phase I, single-center, randomized, open-label, single-dose, 2-way, 2-period, crossover study to evaluate the effect of food on the pharmacokinetics (PK) of vamifeport prolonged-release (PR) formulation in healthy adult participants. Participants will be randomly allocated to one of two treatment sequences.

ELIGIBILITY:
Inclusion Criteria:

* •Aged greater than or equal to (>=) 18 to less than or equal to (<=) 60 years at the time of providing written informed consent.
* •Healthy, as determined by the investigator based on review of defined assessments during Screening.
* •Body weight between 50 and 100 kilogram (kg) (inclusive) and body mass index within the range 18.0 to 30.0 kg per square metre (kg/m2) (inclusive) at Screening and Day - 1.

Exclusion Criteria:

* •Any clinically relevant abnormal means of triplicate 12-lead ECG finding at Screening or Day - 1 (as deemed by the investigator).
* •Serum ferritin of less than (<) 30 nanograms per milliliter (ng/mL) or greater than (>) 300 ng/mL for assigned male at birth (AMAB) participants or < 16 ng/mL or > 300 ng/mL for assigned female at birth (AFAB) participants at Screening or Day - 1.
* •Hemoglobin < 13 gram per deciliter (g/dL) (8.1 millimole per liter [mmol/L]) for AMAB participants or < 12 g/dL (7.5 mmol/L) for AFAB participants at Screening or Day - 1.
* •Blood draw or donation of blood (>= 450 mL) within 3 months before Screening, plasma donation from 2 weeks before Screening, or platelet donation from 6 weeks before Screening.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2025-05-27 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-04 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration (AUC0-last) of vamifeport | 0-96 hours after dose
AUC from time zero extrapolated to infinity (AUC0-inf) of vamifeport | 0-96 hours after dose
Maximum observed plasma concentration (Cmax) of vamifeport | 0-96 hours after dose

SECONDARY OUTCOMES:
Number of participants with treatment emergent adverse events (TEAEs) overall, by severity, seriousness, and relationship to vamifeport | Up to Day 13 (+/- 2 days)
Percentage of participants with TEAEs overall, by severity, seriousness, and relationship to vamifeport | Up to Day 13 (+/- 2 days)
Number of participants with clinically significant changes from baseline in clinical laboratory safety tests (biochemistry, hematology, and urinalysis), 12-lead electrocardiogram (ECG), and vital signs, reported as TEAEs | Up to Day 13 (+/- 2 days)
Percentage of participants with clinically significant changes from baseline in clinical laboratory safety tests (biochemistry, hematology, and urinalysis), 12-lead ECG, and vital signs, reported as TEAEs | Up to Day 13 (+/- 2 days)
Time of the maximum observed plasma concentration (Tmax) of vamifeport | 0-96 hours after dose
Apparent terminal disposition phase plasma half life (t1/2) of vamifeport | 0-96 hours after dose
Apparent terminal disposition rate constant (λz) of vamifeport | 0-96 hours after dose
Apparent total clearance (CL/F) of vamifeport | 0-96 hours after dose
Apparent volume of distribution (V/F) of vamifeport | 0-96 hours after dose
Percentage of AUC due to extrapolation from the last quantifiable concentration to infinity (%AUCextrap) of vamifeport | 0-96 hours after dose
Time of the last quantifiable concentration (Tlast) of vamifeport | 0-96 hours after dose
The time taken for vamifeport to appear in the systemic circulation following administration (Tlag), when applicable | 0-96 hours after dose
AUC from time zero to 12 hours (AUC0-12) and 24 hours (AUC0-24) of vamifeport | 0-12 hours post-dose and 0-24 hours after dose
Plasma concentration of vamifeport | At 12 hours and 24 hours after dose

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring
Locations (1):
- Investigator Site 82600083, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider on a case-by-case basis requests to share Individual Patient Data (IPD) with external bona-fide, qualified scientific and medical researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
Supporting Information: Study Protocol, SAP
Access Criteria: Proposed research should seek to answer a previously unanswered important medical or scientific question.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.